CLINICAL TRIAL: NCT02493907
Title: A Prospective Clinical Trial of Corrected Left Ventricular Electrical Delay Predicting Response to Cardiac Resynchronization Therapy in Chinese With Heart Failure
Brief Title: Corrected Left Ventricular Electrical Delay Predicting Response to Cardiac Resynchronization Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Southern Medical University, China (Other); Fudan University (Other); Beijing Chao Yang Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingfeng Wang, subdecanal, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: [2014] ethics register [34]
Record Dates: First submitted 2015-07-02; First posted 2015-07-10 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Chronic Heart Failure; Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- heart failure: heart failure patients with CRT

SUMMARY:
Cardiac resynchronization therapy (CRT) is a well-established treatment for patients with severe systolic heart failure (HF) and ventricular desynchronization. Despite the consistently observed structural and functional improvements as well as reductions in HF events and mortality in large multicenter randomized trials, 30% patients remain classified as nonresponders. Present evidences showed that QRS duration was the most effective parameter to predict responsivity of CRT in patients with severe HF. But some studies showed that QRS duration could be influenced by obesity and gender. Accordingly, the simple QRS interval width of body surface electrocardiograph should not be the most satisfactory parameter for screening patients suitable for CRT. Recent study showed that left ventricular electrical delay, as measured by the time from the onset of QRS to the LV electrogram peak (QLV), predicted CRT response. At long QLV intervals, atrioventricular optimization (AVO) can increase the likelihood of structural response to CRT. However, it is unclear whether it is suitable for Chinese patients. The investigators would like to validate this relation in a Chinese population and explore if a corrected QLV might do better to predict the responsivity of CRT.

ELIGIBILITY:
Inclusion Criteria:

* •More than 18 Years

  * Informed consent signed
  * NYHA class ≥ II, an ejection fraction of ≤ 0.35, QRS duration of ≥ 150 milliseconds with Non-LBBB) or ≥ 120 milliseconds with LBBB, who treated with CRT
  * The Estimated survival time was more than one year
  * sinus rhythm, pacemaker independent

Exclusion Criteria:

* •NYHA class I symptoms

  * Severe liver or kidney dysfunction
  * Valvular heart disease
  * Pregnancy or lactation women
  * percutaneous coronary intervention (PCI) or cardiac artery bypass graft (CABG) within 3 month
  * Have malignant tumors and the Estimated survival time was less than one year
  * an enzyme-positive myocardial infarction within 3 months before enrollment, or atrial fibrillation
  * any reasons cannot complete follow-up; Or researchers think that don't suit to be included in the research of other conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients received CRT in Sun Yat-sen Memorial Hospital, Sun Yat-sen University. Informed consent must be obtained for all of the included patients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular End Systolic Volume (LVESV) | baseline and 6 months
  change in LVESV

SECONDARY OUTCOMES:
New York Heart Association (NYHA) | baseline and 6 months
  change in NYHA
left ventricular ejection fraction (LVEF) | baseline and 6 months
  change in LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Jingfeng Wang, M.D., Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China